CLINICAL TRIAL: NCT03187379
Title: Efficacy of Exparel (TM) on Post-operative Pain After Laparoscopic Gastric Bypass Using Circular EEA Stapler
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Matthew Kroh (Other)
Responsible Party: Sponsor-Investigator, Matthew Kroh, Principal investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1571
Record Dates: First submitted 2017-06-01; First posted 2017-06-14 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Post-operative Pain Management
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel, Liposomal Bupivacaine (Experimental): Subjects in this arm will receive Exparel® liposomal bupivacaine injected concurrently with 0.25% bupivacaine at the incisional sites prior to closing
  Interventions: Drug: Exparel
- Control (Active Comparator): Subjects in this arm will receive 0.25% bupivacaine alone
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel — Exparel liposomal bupivacaine - 20cc Exparel® + 60cc Bupivicaine
  Arms: Exparel, Liposomal Bupivacaine
Drug: Bupivacaine — 60cc Bupivacaine
  Arms: Control

SUMMARY:
This will be a comparative study between two cohorts of patients undergoing Roux-en-Y Gastric bypass. One cohort (75 patients) will receive FDA approved Exparel® (liposome bupivacaine injection solution) injections intra-operatively at time of incision site closure. The control cohort (75 patients) will receive 0.25% bupivacaine injection solution at the time of incision site closure. The medication for the control group is our current standard of care. The primary end point is post-operative pain at 24 and 48 hours measured by the Visual Analog Scale (VAS). Comparison will be made between cohorts. All subjects enrolled in the study will be evaluated per nursing protocol with the verbal numerical analog scale. At 24 and 48 hours a member of the research team will administer a 2-part questionnaire containing the VAS and the Revised American Pain Society Post-Operative Questionnaire (APS-POQ-R). The latter is validated for assessment of the patient's experience of pain and it hindrance to daily activity in the post operative period.

DETAILED DESCRIPTION:
The study will include up to 150 patients, and will consist of two cohort. The study cohort will include 75 patients who receive intraoperative Exparel® injections at the incision locations in addition to our standard multimodality post-operative analgesia. The control arm will include 75 patients who meet inclusion criteria but receive standard 0.25% bupivacaine and our standard multimodality post-operative analgesia. Patients will be randomized by REDCap™ database system in collaboration with Cleveland Clinic Pharmacy to receive either Exparel® or the control medication (0.25% Bupivacaine). Consent from patients will be obtained and documented by a dedicated research personnel prior to any enrollment.

ELIGIBILITY:
Inclusion Criteria:

* bariatric surgery patients
* laparoscopic roux-en-y gastric bypass
* use of EEA stapler anastomosis

Exclusion Criteria:

* age <18 years
* previous history of roux-en-y gastric bypass
* patients undergoing other bariatric procedures
* pre-operative opioid analgesics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alisan Fathalizadeh, M.D, Principal Investigator — Staff
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel, Liposomal Bupivacaine | Control
Started | 50 | 52
Completed | 50 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel, Liposomal Bupivacaine | Control | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 48.4 [37.1 to 56.2] | 41.2 [36.3 to 52.2] | 44.6 [36.7 to 55.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Pain
Description: Patient-reported pain levels, on a 0-100 Visual Analog Scale (VAS) with 0 representing less pain and 100 representing more pain.
Time Frame: 24 hours post-surgery
Measure: Mean (Standard Deviation); unit: units on a Visual Analog Scale (VAS)
Arm/Group | Exparel, Liposomal Bupivacaine | Control
Number analyzed (Participants) | 50 | 52
units on a Visual Analog Scale (VAS) | 49.4 (29) | 56.6 (26.4)

2. Secondary Outcome: Post-Operative Pain
Description: as for outcome 1
Time Frame: 48 hours post-surgery
Measure: Mean (Standard Deviation); unit: units on a Visual Analog Scale (VAS)
Arm/Group | Exparel, Liposomal Bupivacaine | Control
Number analyzed (Participants) | 50 | 52
units on a Visual Analog Scale (VAS) | 42.2 (30) | 51.5 (31.4)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Exparel, Liposomal Bupivacaine | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 10/50 | 15/52
Other Adverse Events (participants affected / at risk) | 14/50 | 27/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel, Liposomal Bupivacaine (N=50) | Control (N=52)
Nausea (General disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
Abdominal Pain (General disorders) | 2 (2) | 5 (5)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Left Side Pain (General disorders) | 0 (0) | 1 (1)
Right Flank Pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Post Operative Complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exparel, Liposomal Bupivacaine (N=50) | Control (N=52)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 3 (3) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4)
Pain- Not otherwise Specified (General disorders) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Wound Drainage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chest Pain (General disorders) | 4 (4) | 2 (2)
Pelvic Pain (General disorders) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Vaginal Bleed (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Leg Burn (General disorders) | 0 (0) | 1 (1)
Left Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dehydration (General disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Abnormal labs (Investigations) | 0 (0) | 1 (1)
Black Stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 2 (2)
Left Side Pain (General disorders) | 1 (1) | 0 (0)
Swollen Leg (General disorders) | 1 (1) | 0 (0)
Right Eye Complaint (Eye disorders) | 0 (0) | 1 (1)
Infection- Not otherwise Specified (Infections and infestations) | 0 (0) | 1 (1)
Hip Pain (General disorders) | 0 (0) | 1 (1)
Congestion (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03187379/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03187379/ICF_001.pdf